CLINICAL TRIAL: NCT02098681
Title: Society for Pediatric Anesthesia Improvement Network (SPAIN) Chest Wall Deformity Project (Pectus Repair)
Brief Title: SPAIN Chest Wall Deformity Project (Pectus Repair)
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other); Children's Hospital Colorado (Other); Children's Hospital Los Angeles (Other); Children's Hospital of Philadelphia (Other); Dartmouth-Hitchcock Medical Center (Other); Alfred I. duPont Hospital for Children (Other); Emory University (Other); Johns Hopkins University (Other); Mayo Clinic (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Joseph P. Cravero, Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00010229
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Deformity of Chest Wall
Keywords: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Context: Chest wall deformities in children are relatively common. One such deformity, known as Pectus Excavatum (PE), involves a concavity of the chest and is the most frequent of these abnormalities - present in approximately 1 out of every 400-1000 births. This deformity is often a cosmetic problem for affected individuals. When severe, PE can also be associated with cardiopulmonary compromise.

Treatment of PE involves surgical correction. There are several potential methods for correcting PE. In the past the most common repair involved an open procedure which involves excision and reshaping of the ribcage. More recently a minimally invasive procedure has been adopted involving the placement of a stainless steel or titanium bar underneath the sternum to reshape the chest wall. This procedure, commonly known as the Nuss procedure, carries with it significant post-operative pain management problems. In fact, the pain issues after Nuss procedure may be more significant than after open repair. The quality of postoperative pain control in these cases has been shown to affect several measurable objective outcomes during hospitalization including capacity for deep breathing, early mobilization, ambulation, and length of hospital stay.

Epidural analgesia (EA) has been one of the standard methods for managing pain in the early postoperative period after PE repair. Unfortunately severe pain may persist after the removal of an epidural catheter resulting in a difficult "transition" period just prior to discharge from the hospital. In addition reports of neurological injury after epidural analgesia for Nuss procedures have appeared. In light of these issues, many institutions have opted for alternative methods of pain control including peripheral nerve blocks, patient controlled analgesia, and wound catheters.

There remains significant debate as to which pain control methodology is best. There is little consistent data available on pain control or outcomes that occur after EA is stopped. Moreover there is reluctance in any one institution to trial or randomize patients to a variety of treatment modalities. For all of these reasons, investigators are proposing participation in a multi-institutional data sharing project concerning the repair of EA in which participating centers will collaborate to better understand the outcomes of perioperative care for patients undergoing correction of this problem.

DETAILED DESCRIPTION:
Context: Chest wall deformities in children are relatively common. One such deformity, known as Pectus Excavatum (PE), involves a concavity of the chest and is the most frequent of these abnormalities - present in approximately 1 out of every 400-1000births. This deformity is often a cosmetic problem for affected individuals. When severe, PE can also be associated with cardiopulmonary compromise.

Treatment of PE involves surgical correction. There are several potential methods for correcting PE. In the past the most common repair involved an open procedure which involves excision and reshaping of the ribcage. More recently a minimally invasive procedure has been adopted involving the placement of a stainless steel or titanium bar underneath the sternum to reshape the chest wall. This procedure, commonly known as the Nuss procedure, carries with it significant post-operative pain management problems. In fact the pain issues after Nuss procedure may be more significant than after open repair. The quality of postoperative pain control in these cases has been shown to affect several measurable objective outcomes during hospitalization including capacity for deep breathing, early mobilization, ambulation, and length of hospital stay.

Epidural analgesia (EA) has been one of the standard methods for managing pain in the early postoperative period after PE repair. Unfortunately severe pain may persist after the removal of an epidural catheter resulting in a difficult "transition" period just prior to discharge from the hospital. In addition reports of neurological injury after epidural analgesia for Nuss procedures have appeared. In light of these issues, many institutions have opted for alternative methods of pain control including peripheral nerve blocks, patient controlled analgesia, and wound catheters. There remains significant debate as to which pain control methodology is best. There is little consistent data available on pain control or outcomes that occur after EA is stopped. Moreover there is reluctance in any one institution to trial or randomize patients to a variety of treatment modalities. For all of these reasons, investigators are proposing participation in a multi-institutional data sharing project concerning the repair of EA in which participating centers will collaborate to better understand the outcomes of perioperative care for patients undergoing correction of this problem.

The primary objective is to create a multicenter registry which captures data relating to the perioperative course and management of children undergoing PE repair surgery. This effort is undertaken in order to augment safety and quality improvement activities at participating sites. Investigators understand that there are multiple methodologies for accomplishing the anesthesia and perioperative pain control for this surgery. There is little comparative data on the outcomes from the different possible management strategies. Given the relative frequencies of these surgeries where few centers perform more than 20-50 of these procedures per year, it is not practical for any one (or two) centers to study this procedure in an observational manner or a controlled randomized trial. Investigators' aggregate multi-institutional data set will be used for benchmarking for both local and national safety and quality improvement efforts. Participating sites will be provided with reports comparing the local site to the aggregate dataset for specific perioperative outcome variables (e.g. pain metrics) and factors that could be associated with improved outcomes. Outcome variables include but are not limited to intraoperative hemodynamics, pain control, emergence agitation, apnea/airway obstruction, hemodynamic stability, time to first ambulation, pain scores while in the hospital, total hospital days, time to school or work attendance, and symptoms of post-traumatic stress.

Secondary objective: Investigators will ultimately look at the relationship between specific management metrics such as the use of epidural anesthesia vs. peripheral nerve blocks vs. local anesthesia wound infiltration and our primary outcome metrics. In addition Investigators will consider the frequency of long term Post Traumatic Stress behaviors and the various measures of pain control in the perioperative period.

Study Design:

Basic design: Prospective observational multicenter data registry

Setting/Participants:

* Patients ages 8 to 30 years undergoing surgery for Pectus Excavatum Repair in a hospital setting
* Up to 20 hospital sites

Data Collection, Storage and Release:

The registry will capture data relating to the perioperative management of children undergoing PE repair. Measures will include demographic data, data on degree of deformity, perioperative management, intraoperative management, hospital course, surgical technique, complications, and long term pain/psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 8 to 30 years.
* Undergoing surgical procedures on the chest wall region performed to correct Pectus Excavatum deformities.

Exclusion Criteria:

* None.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals undergoing surgical procedures on the chest wall region performed to correct Pectus Excavatum deformities.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10-20 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline, Daily up to Three Weeks
  Peri- and Post-Operative Pain Control

SECONDARY OUTCOMES:
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline
  Intraoperative Hemodynamics
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline
  Emergence Agitation
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline
  Apnea/Airway Obstruction
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline
  Hemodynamic Stability
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline, up to Three Weeks
  Time to First Ambulation
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline, until Discharge From Hospital (Up to Three Weeks)
  Pain Scores
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Baseline, until Discharge from Hospital (Up to Three Weeks)
  Total Hospital Days
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Up To Three Months After Hospital Discharge
  Time to School or Work Return
Perioperative course and management of children undergoing Pectus Excavatum repair surgery. | Up to Three Months After Hospital Discharge
  Symptoms of Post-Traumatic Stress

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Cravero, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States